CLINICAL TRIAL: NCT04631406
Title: A Phase 1/Phase 2a Safety and Tolerability Study of Intracerebral Transplantation of Neural Stem Cells (NR1) in Subjects With Chronic Ischemic Subcortical Stroke (ISS) and Early Evaluation of Potentially Useful Efficacy Parameters
Brief Title: A Safety and Tolerability Study of Neural Stem Cells (NR1) in Subjects With Chronic Ischemic Subcortical Stroke (ISS)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gary Steinberg, MD, PhD (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor-Investigator, Gary Steinberg, MD, PhD, Professor and Former Chair, Department of Neurosurgery, School of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NR1-02
Record Dates: First submitted 2019-04-11; First posted 2020-11-17 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neural Stem cells injected intracerebrally (Experimental): Subject cohorts will be treated with increasing doses of Neural Stem Cells injected intracerebrally using a traditional 3+3 trial design
  Interventions: Biological: Neural Stem Cells

INTERVENTIONS:
Biological: Neural Stem Cells — NR1 is a human embryonic stem cell (hESC) derived product for the treatment of chronic ischemic subcortical stroke

SUMMARY:
Evaluation of the safety and tolerability of escalating doses of NR1 administered intracerebrally at a single time-point post-injury to subjects with chronic ISS with or without cortical stroke.

DETAILED DESCRIPTION:
Evaluation of the safety and tolerability of escalating doses of NR1 administered intracerebrally at a single time-point post-injury to subjects with chronic ISS with or without cortical stroke. The study will be a dose escalation using up to 4 cohorts each at a single dose level, of intracerebral administration of NR1 cells. Secondary objectives are to evaluate clinical and radiologic responses as well as utility of efficacy measurement tools.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* History of ischemic subcortical stroke in the middle cerebral artery and/or lenticulostriate artery 6 to 60 months from time of stroke
* Ability of subject to understand and provide written Informed Consent
* Willing to take tacrolimus (Prograf) 2 days before and for 2 months after transplant

Exclusion Criteria:

* Stroke lesion less than 1 cubic centimeter or greater than 100 cubic centimeters measured by MRI
* Index stroke is lacunar infarct less than 1 year old
* History or presence of any major neurological disease
* History of active cancer other than basal or squamous cell skin cancers
* History of seizures
* Pregnant or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 0-12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Fugl Meyer (FM) motor score | 0-12 months
  Change in neurologic functional outcome to evaluate efficacy post-injection as defined by change in Fugl Meyer motor score in comparison to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gary K Steinberg, MD, PhD, Principal Investigator — Professor, Neurosurgery Department
Locations (1):
- Stanford Health Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No